CLINICAL TRIAL: NCT05596032
Title: Prospective Field Study to Validate the Diagnostic Performance of the IVD CAPSULE COVID-19-NP Test for the Detection of SARS-CoV-2 on abioSCOPE®
Brief Title: Prospective Study to Validate the Diagnostic Performance of IVD CAPSULE COVID-19-NP Test for the Detection of SARS-CoV-2
Status: Completed | Type: Observational
Sponsor: Abionic SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-COV-003
Record Dates: First submitted 2022-10-21; First posted 2022-10-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to conduct a prospective evaluation of the diagnostic performance of the IVD CAPSULE COVID-19-NP test for antigenic determination of SARS-CoV-2 virus on the abioSCOPE® instrument.

The objective of the clinical study is to demonstrate that the IVD CAPSULE COVID-19-NP test:

1. shows sensitivity:

   * ≥ 80% when testing unselected symptomatic participants within the first seven days of symptom onset or asymptomatic participants when diagnosis is confirmed by RT-PCR; Or
   * ≥ 90% for subjects with Ct ≤ 25.
2. show ≥ 98% specificity.

ELIGIBILITY:
Inclusion Criteria:

* provide valid informed consent before taking the tests;
* in the case of symptomatic patients, be tested within the first seven days after the onset of symptoms.
* Male or female, aged equal to or older than 18 years of age.

Exclusion Criteria:

* Symptomatic participants who take the test after seven days after the onset of symptoms are excluded from the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes unselected participants*, symptomatic, asymptomatic having had close contact with positive patients, and asymptomatic with no known exposure to SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2022-10-23 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of the IVD CAPSULE COVID-19-NP antigenic test | through study completion, an average of 1 month
  The purpose of this work is to carry out a prospective evaluation of the diagnostic performance of the IVD CAPSULE COVID-19-NP test for the antigenic determination of the SARS-CoV-2 virus on the abioSCOPE instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- A.O Mauriziano di Torino, Torino, Italy